CLINICAL TRIAL: NCT06057571
Title: A Phase II, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Oral TT-00420 (Tinengotinib) Tablets in Subjects With Cholangiocarcinoma Who Failed or Relapsed to Prior Treatment of Chemotherapy and FGFR Inhibitor
Brief Title: Study of TT-00420 (Tinengotinib) in Subjects With Cholangiocarcinoma Who Failed or Relapsed to Chemotherapy and FGFR Inhibitor
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT00420CN08
Record Dates: First submitted 2023-09-05; First posted 2023-09-28 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cholangiocarcinoma Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TT-00420 (tinengotinib) Tablet Monotherapy (Experimental): TT-00420 (tinengotinib) tablets will be administered once daily in 21-day cycles with initial dosage of 10 mg QD.
  Interventions: Drug: TT-00420 (tinengotinib)

INTERVENTIONS:
Drug: TT-00420 (tinengotinib) — TT-00420 (tinengotinib) tablet will be administered orally once daily per protocol defined schedule.

SUMMARY:
A phase II, open-label, multicenter study to evaluate the efficacy and safety of oral TT-00420 (Tinengotinib) tablets in subjects with cholangiocarcinoma who failed or relapsed to prior treatment of chemotherapy and FGFR Inhibitor.

DETAILED DESCRIPTION:
Approximately 50 subjects will be enrolled. Eligible subjects will receive tinengotinib 10 mg QD orally as the initial dose level in 21-day cycles until confirmed disease progression, intolerable toxicity, death, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Histologically or cytologically confirmed CCA/adenocarcinoma of biliary origin with radiological evidence of unresectable or metastatic disease.
3. Subjects must have received one or two lines of prior systemic chemotherapy.
4. Documentation of FGFR2 gene alteration and must have failed to prior treatment of exactly one FGFR inhibitor.
5. At least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors.
6. ECOG≤ 1.
7. Adequate organ and bone marrow function(without receiving any hematopoietic growth factor, blood or platelet therapy within 14 days before the first dose).
8. Must agree to take sufficient contraceptive methods to avoid pregnancy during the study and until at least 3 months after ceasing study treatment.
9. Able to sign informed consent and comply with the protocol.

Exclusion Criteria:

1. Subjects with concomitant brain or central nervous system (CNS) metastases and imaging or clinically confirmed progression within 28 days prior to the start of treatment. Brain or central nervous system metastases that not treated with corticosteroids and remain stable within 14 days prior to screening are eligible for enrollment.
2. Subjects with a known concurrent malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, including those that have previously undergone potentially curative therapy.
3. Subjects who have received prior systemic therapy or investigational study drug ≤ 5 half-lives or 14 days, whichever is shorter, prior to starting the study drug or who have not recovered (grade ≤ 1 or at pretreatment baseline except tolerable grade 2 alopecia, fatigue/asthenia, and neuropathy due to trauma) from adverse events (AEs) of prior therapy.
4. Concurrent anticancer therapy including chemo-, immune-, or radiotherapy. Hormone therapy may be allowed with Sponsor approval.
5. Subjects who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting the study drug or who have not recovered from AEs of prior therapy.
6. Subjects who have underwent major surgery or have not recovered from adverse events of surgery within the 4 weeks prior to initiation of the investigational drug (grade ≤ 1 or at pretreatment baseline except tolerable grade 2 alopecia, fatigue/asthenia, and neuropathy due to trauma).
7. Impaired cardiac function or significant diseases.
8. Subjects who have received stable doses of antihypertensive drugs for at least 1 week with uncontrolled hypertension under at screening period (defined as blood pressure of ≥ 150 mm Hg systolic and/or ≥ 90 mm Hg diastolic despite adequate treatment with antihypertensive medications at screening).
9. Subjects who have severe gastrointestinal disease or gastrointestinal dysfunction that may lead to absorption, metabolism or excretion of the study drug, enrollment eligibility will be based on the investigator's judgment (including but not limited to total gastrotomy, short bowel syndrome).
10. Subjects who have bleeding disorders or thrombotic disorders or therapeutic anticoagulant therapy requiring INR monitoring.
11. Subjects who have received a strong CYP3A inhibitor and inducer before starting the study drug, within an interval of ≤ 2 weeks or 5 half-lives (whichever is shorter); (except topical ketoconazole).
12. Tested positive for the human immunodeficiency virus (HIV).
13. Subjects who have an active HBV infection.
14. Subjects who are pregnant or breastfeeding.
15. Subjects who are unable to swallow or tolerate oral medication.
16. The investigator determines that he or she is not eligible for study participation for any clinical or laboratory abnormalities, or any reason that could confuse the study results, interfere with participants' safe participation and compliance with the trial procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by BICR | Through study completion, an average of 1 year
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, an average of 1 year
  From first study drug administration until the date of first documented progression or date of death from any cause, whichever came first
Overall Survival (OS) | Through study completion, an average of 1 year
  From first study drug administration until the date of death from any cause
ORR by Investigator | Through study completion, an average of 1 year
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.
Disease control rate (DCR) | Through study completion, an average of 1 year
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) or a stable disease (SD) based on RECIST version 1.1.
Duration of response (DOR) | Through study completion, an average of 1 year
  Duration of response for CR or PR based on RECIST version 1.1.
Incidence, duration, and severity of adverse events (AEs) | Up to 28 days from study discontinuation
  As assessed per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (or the most current version).

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Qianhai Shekou Free Trade Zone hospital, Shenzhen, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Zhongnan hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Central Hospital Affiliated to Shangdong First Medical University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Beijing Tsinghua Changgeng Hospital, Beijing
  - Fudan University Shanghai Cancer Hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - Tianjin medical university cancer institute & hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No